CLINICAL TRIAL: NCT06999369
Title: Heart Failure Food Intervention Trial (HF-FIT): Impact of a Guideline-based Nutrition Digital Tool in Heart Failure Patient Clinical Outcomes
Brief Title: Heart Failure Food Intervention Trial: Impact of a Guideline-based Nutrition Digital Tool in Heart Failure Patient Clinical Outcomes
Acronym: HF-FIT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sutter Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024.112EXP; 382101125-0525 (Other: Sutter Health)
Record Dates: First submitted 2025-05-14; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
Keywords: heart failure; nutrition app; evidence-based nutrition recommendations; guideline-based nutrition app; app-based dietary intervention
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Patients in the control arm will be asked to complete a baseline survey questionnaire and a final survey questionnaire 6 months after they enroll. During enrollment or (if not obtained at baseline) up to 1 month after, patients will be asked to provide their baseline BP and weight measurements. Study team members will contact patients at month 3 and 6 to ask how they are doing and get follow up BP and weight measurements.
- Intervention: MedChefs (Experimental): Once patients have been randomized to the MedChefs arm, they will be contacted by the research team and sent an email link to use the MedChefs app During enrollment or up to 1 month after, patients will be contacted to provide their baseline BP and weight measurements. Patients will be contacted at month 3 and 6 by the research team to see how they are doing, about their app use, get their BP and weight measurements and will be sent a final survey 6 months after they first log into MedChefs.
  Interventions: Other: MedChef App
- MedChefs plus Instacart Food Voucher (Experimental): Once patients have been randomized to the MedChefs arm and voucher arm, they will be contacted by the research team and sent an email link to use the MedChefs app. Patients will also be given a $100 voucher to buy food recommended by the app. Vouchers will be provided once a month for the 6 months of the study. During enrollment or up to 1 month after, patients will be asked to provide their baseline BP and weight measurements. At month 3 and 6 the research team will contact the patients to see how they are doing and ask for patients follow up BP and weight measurements. Patients will also be asked to complete a final survey 6 months after they first log into MedChefs.
  Interventions: Other: MedChef App; Other: MedChefs and Instacart food voucher

INTERVENTIONS:
Other: MedChef App — Once patients have been randomized to the MedChefs arm, they will be contacted by the research team and sent an email link to use the MedChefs app. The research team will contact the patient based on their preferred contact method and will walk through how to use the app and share education on its use.
  Other Names: Nutritional App
  Arms: Intervention: MedChefs; MedChefs plus Instacart Food Voucher
Other: MedChefs and Instacart food voucher — Once patients have been randomized to the MedChefs arm and voucher arm, they will be contacted by the research team and sent an email link to use the MedChefs app. The research team will contact the patient based on their preferred contact method and will walk through how to use the app and share education on its use and use of Instacart food vouchers. Patients will also be given a $100 voucher to buy food recommended by the app. Vouchers will be provided once a month for the 6 months of the study
  Other Names: nutrition app; food voucher
  Arms: MedChefs plus Instacart Food Voucher

SUMMARY:
Measuring the impact of a guideline-based nutrition digital tool in heart failure patients

DETAILED DESCRIPTION:
The goal of this research clinical trial is to learn understand or learn whether a guideline-based nutrition application (app) called MedChefs can help heart failure patients adopt and sustain an evidence-based dietary patterns.

ELIGIBILITY:
Inclusion Criteria:

* 18-89 years old at time of enrollment
* Any type of Heart failure diagnosis (e.g., I50.x) between 1/1/2023-present
* Recent hospital admission (within a year)
* Race/ethnicity: All race/ethnic groups
* Location: patients have been treated in the Greater East Bay division and Greater Silicon Valley division areas.
* Patients with have at least 1 office/outpatient visit with a primary care physician or cardiologist visit before index date

Exclusion Criteria:

* • Patients with certain patient history (cognitive disabilities) and end stage renal or metastatic cancer diagnosis

  * Patients with active drug/substance use. Patients with heart failure who have active substance use are excluded from the study. HF patients with substance use require additional monitoring and follow up due to potential severe withdrawal symptoms, acute HF exacerbation and drug overdose or medication errors. Standard protocol includes additional monitor vital signs (e.g., blood pressure, heart rate) and HF symptoms (e.g., edema, dyspnea), and performing regular laboratory tests (e.g., renal function, electrolytes) which is beyond the clinical and logistical capabilities of this study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Baseline and 6 months
  Blood pleasure will be measure by mmHg

SECONDARY OUTCOMES:
Weight | Baseline and 6 months
  Weight will be measured in pounds

CONTACTS AND LOCATIONS:
Locations (1):
- 2121 N. California Blvd., Suite 310, Walnut Creek, California, United States

IPD SHARING:
Plan to Share IPD: No